CLINICAL TRIAL: NCT02013700
Title: A Phase I, Randomized, Blinded and Placebo-controlled Trial to Evaluate the Safety, Tolerability, and Potential Efficacy of Allogeneic Human Mesenchymal Stem Cell Infusion in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Allogeneic Human Cells (hMSC)in Patients With Idiopathic Pulmonary Fibrosis Via Intravenous Delivery (AETHER)
Acronym: AETHER
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study completed
Sponsor: Joshua M Hare (Other)
Collaborators: The Lester And Sue Smith Foundation (Unknown); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor-Investigator, Joshua M Hare, Chief Science Officer / Director of Interdisciplinary Stem Cell Institute, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20120946
Record Dates: First submitted 2013-12-02; First posted 2013-12-17 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
Keywords: IPF; Pulmonary fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 20 million hMSCs (Experimental): Patients will receive a single administration of Allogeneic Adult Human Mesenchymal Stem Cells (hMSCs): 2 x10^6 (20 million) cells delivered via peripheral intravenous infusion
  Interventions: Biological: Allogeneic Adult Human Mesenchymal Stem Cells (hMSCs)
- Placebo (Placebo Comparator): Patients will receive a matched placebo delivered via peripheral intravenous infusion
  Interventions: Biological: matched placebo
- 100 million hMSCs (Experimental): Patients will receive a single administration of Allogeneic Adult Human Mesenchymal Stem Cells (hMSCs): 100 x10^6 (20 million) cells delivered via peripheral intravenous infusion
  Interventions: Biological: Allogeneic Adult Human Mesenchymal Stem Cells (hMSCs)
- 200 million hMSCs (Experimental): Patients will receive a single administration of Allogeneic Adult Human Mesenchymal Stem Cells (hMSCs): 200 x10^6 (200 million) cells delivered via peripheral intravenous infusion
  Interventions: Biological: Allogeneic Adult Human Mesenchymal Stem Cells (hMSCs)

INTERVENTIONS:
Biological: Allogeneic Adult Human Mesenchymal Stem Cells (hMSCs)
  Arms: 100 million hMSCs; 20 million hMSCs; 200 million hMSCs
Biological: matched placebo — The placebo will be 25 ml of Plasma-Lyte A with 1% HSA in a Cryostore bag.
  Arms: Placebo

SUMMARY:
This is a phase I, randomized, blinded, placebo-controlled 9 subjects pilot safety run-in followed by an additional 16 randomized subjects for a total of 25 subjects. In the pilot phase subjects will be randomized into three treatment groups of allogenic mesenchymal stem cells and in the randomized phase subjects will receive either allogenic mesenchymal stem cells or matched placebo.

DETAILED DESCRIPTION:
Idiopathic Pulmonary Fibrosis (IPF) is a progressive and debilitating lung disease characterized by interstitial fibrosis with decreasing lung volumes and pulmonary insufficiency eventually resulting in death. Patients with Idiopathic Pulmonary Fibrosis (IPF) typically present with complaints of sub acutely progressive dyspnea and non-productive cough, often accompanied by digital clubbing. Due to the insidious onset of symptoms, however, most patients are diagnosed at late stages of the disease after significant fibrosis has occurred. Physical exam is characterized by hypoxemia, "dry" inspiratory crackles on auscultation, and occasional digital clubbing (6). Pulmonary function tests (PFTs) usually reveal restrictive lung physiology with progressive decline of forced vital capacity (FVC), diffusion capacity (DLCO) and six-minute walk distances. Diagnosis is established by the pathologic finding of usual interstitial pneumonia (with sub epithelial fibroblastic foci) by open lung biopsy (7), and/or by high resolution CT (HRCT) demonstrating the characteristic findings of peripheral/basal sub pleural reticulonodular changes with fibrosis, honeycombing, and traction bronchiectasis (8, 9).

The prognosis for patients with Idiopathic Pulmonary Fibrosis (IPF) is uniformly poor. The natural history of the disease is characterized by inexorable progressive decline interspersed with "exacerbations" or periods of accelerated disease which are often fatal (5). There are no FDA approved treatment options for patients with Idiopathic Pulmonary Fibrosis (IPF) and thus no standard of care. In cases of patients under the age of 60 with limited comorbid disease, lung transplant may be offered. Patients with Idiopathic Pulmonary Fibrosis (IPF) receive empiric treatment, supportive care alone, and more recently, are offered enrollment in clinical trials.

The pathogenesis of Idiopathic Pulmonary Fibrosis (IPF) is characterized by epithelial cell injury and activation with interstitial inflammation, fibroblast proliferation with extracellular matrix collagen deposition, and eventual loss of function. Because mesenchymal stem cells are known to home to sites of injury, inhibit inflammation, and contribute to epithelial tissue repair, their use has been suggested as a novel therapy for the treatment of Idiopathic Pulmonary Fibrosis (IPF).

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent.
* Subjects age equal to or greater than 40 and equal to or less than 90 years at the time of signing the Informed Consent Form.
* Have a clinical diagnosis of Idiopathic Pulmonary Fibrosis (IPF) prior to screening
* Forced vital capacity (FVC) ≥ 50% predicted and diffusing capacity (DLCO) ≥30% (corrected for hemoglobin but not alveolar volume).
* RVSP equal to or less than 50 mmHg, as documented by Doppler echo or right heart catheterization.
* Female subjects must be surgically sterile or post-menopausal (greater than 1 year).

Exclusion Criteria:

* HRCT and/or surgical lung biopsy results inconsistent with the diagnosis of IPF.
* Infiltrative lung disease of any type other than Idiopathic Pulmonary Fibrosis (IPF), lungs disease related to fibrogenic agents, toxins, drugs or other exposures, granulomatous lung disease, pulmonary vascular disease, or known connective tissue disease.
* Inability to perform any of the assessments required for endpoint analysis (report safety or tolerability concerns, perform pulmonary function tests or high resolution CT (HRCT), undergo blood draws, read and respond to questionnaires.
* Currently receiving (or received within four weeks of screening) any medication, treatment, or experimental agents for the treatment of Idiopathic Pulmonary Fibrosis (IPF), except for patients receiving non drug therapies will include oxygen saturation therapy (oxygen supplementation) and pulmonary rehabilitation.
* Active listing (or expected future listing) for transplant of any organ.
* Clinically important abnormal screening laboratory values, including but not limited to: hemoglobin <8 g/dl, white blood cell count <3000/mm3, platelets <80,000/mm3, INR > 1.5, aspartate transaminase, alanine transaminase, or alkaline phosphatase > 3 times upper limit of normal, total bilirubin > 1.5 mg/dl.
* Serious comorbid illness that, in the opinion of the investigator, may compromise the safety or compliance of the patient or preclude successful completion of the study. Including, but not limited to: HIV, advanced liver or renal failure, class III/IV congestive heart failure, myocardial infarction, unstable angina, or cardiac revascularization within the last six months, or severe obstructive ventilatory defect.
* Any other condition that, in the opinion of the investigator, may compromise the safety or compliance of the patient or preclude successful completion of the study.
* Have known allergies to penicillin or streptomycin.
* Be an organ transplant recipient.
* Have a clinical history of malignancy within 5 years (i.e., patients with prior malignancy must be disease free for 5 years), except curatively- treated basal cell carcinoma, squamous cell carcinoma, or cervical carcinoma.
* Have a non-pulmonary condition that limits lifespan to less than 1 year.
* Have a history of drug or alcohol abuse within the past 24 months.
* Be serum positive for Human immunodeficiency virus (HIV), hepatitis BsAg or Viremic hepatitis C.
* Be currently participating (or participated within the previous 30 days) in an investigational therapeutic or device trial.
* Be a female who is pregnant, nursing, or of childbearing potential while not practicing effective contraceptive methods. Female patients must undergo a blood or urine pregnancy test at screening and within 36 hours prior to injection.
* Female subjects must have a FSH less than 25.8 IU/L
* Subject with hypersensitivity to dimethyl sulfoxide (DMSO)
* Saturated oxygen (SpO2 of less than 93% (room air [sea level] at rest). SpO2 of less than 88% (room air [>5,000 feet above sea level (1524 meters) at rest).

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-11-13 (Actual); Primary Completion 2015-12-11 (Actual); Study Completion 2016-11-24 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of intravenous allo hMSCs in patients with Idiopathic Pulmonary Fibrosis (IPF). | One month post infusion
  Safety (Primary): Incidence (one month post infusion) of any treatment-emergent serious adverse events (TE-SAEs), defined as the composite of: death, non-fatal pulmonary embolism, stroke, hospitalization for worsening dyspnea and clinically significant laboratory test abnormalities.

SECONDARY OUTCOMES:
- To explore effects of allo hMSCs on lung function: forced vital capacity (FVC). | Participants will be followed from 12 weeks to an expected average of 60 weeks following infusion.
  - Difference in absolute decline of forced vital capacity (FVC) percent predicted.
To explore effects of allogenic human mesenchymal stem cells on symptom related quality of life. | Participants will be followed from 4 weeks to an expected average of 60 weeks following infusion.
  - Quality of Life endpoint tools to be used include: University of California San Diego-Shortness of breath (UCSD-SOBQ), short form - 36 (SF-36), and St. George's respiratory questionnaire (SGRQ) questionnaires.
Difference in frequency of acute exacerbations of Idiopathic Pulmonary Fibrosis (IPF) | 4 weeks following infusion
  Defined as:
  * New or worsened dyspnea (<30 days).
  * New ground glass opacities on High Resolution CT (HRCT) superimposed on chronic findings.
  * New or worsened hypoxemia in the absence of other identifiable causes.
Death from any cause. | 60 weeks.
  Participants will be followed for the duration of the trial, which is an expected average of 60 weeks.
To explore effects of allogenic human mesenchymal stem cells on lung function: Diffusing Capacity (DLCO) | Participants will be followed from 12 weeks to an expected average of 60 weeks following infusion.
  - Difference in absolute decline of Diffusing capacity (DLCO).

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn K. Glassberg, MD, Principal Investigator — University of Miami
Locations (1):
- Interdisciplinary Stem Cell Institute / University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Glassberg MK, Minkiewicz J, Toonkel RL, Simonet ES, Rubio GA, DiFede D, Shafazand S, Khan A, Pujol MV, LaRussa VF, Lancaster LH, Rosen GD, Fishman J, Mageto YN, Mendizabal A, Hare JM. Allogeneic Human Mesenchymal Stem Cells in Patients With Idiopathic Pulmonary Fibrosis via Intravenous Delivery (AETHER): A Phase I Safety Clinical Trial. Chest. 2017 May;151(5):971-981. doi: 10.1016/j.chest.2016.10.061. Epub 2016 Nov 24. PMID 27890713
- See also: Interdisciplinary Stem Cell Institute University of Miami — http://isci.med.miami.edu/